CLINICAL TRIAL: NCT05884905
Title: Randomized Study Evaluating Safety of Short Hydration Method for Cisplatin Administration Compared With Conventional Hydration
Brief Title: Safety of Short Hydration Method for Cisplatin Administration Compared With Conventional Hydration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: si186/2023
Record Dates: First submitted 2023-04-30; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Renal Insufficiency; Cis-Platinum Nephropathy
Keywords: renal impairment; cisplatin; hydration protocol
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short hydration (Experimental): Normal saline (NSS) 500 ml infusion in 1 hour cisplatin in NSS 100 ml with 20% mannitol 100 ml infusion in 1 hour other chemotherapy infusion in 1 hour (if available) NSS 500 ml infusion in 1 hour, then NSS 500 ml infusion in 2 hours
  Interventions: Procedure: short hydration
- conventional hydration (Other): NSS 1000 ml infusion in 8 hour cisplatin in NSS 100 ml with 20% mannitol 100 ml infusion in 1 hour other chemotherapy infusion in 1 hour (if available) NSS 2000 ml infusion in 16 hour
  Interventions: Procedure: conventional hydration

INTERVENTIONS:
Procedure: short hydration — NSS infusion prior to and following cisplatin administration within 6 hours
  Other Names: short intravenous fluid infusion
  Arms: short hydration
Procedure: conventional hydration — NSS infusion prior to and following cisplatin administration over 24 hours
  Other Names: long intravenous fluid infusion
  Arms: conventional hydration

SUMMARY:
The aim of the study is to evaluate safety of short hydration with cisplatin administration. The main outcome is renal dysfunction following cisplatin use with short hydration protocol. Another group of patients received conventional hydration is the historical control for comparison (Randomized phase II design with a reference standard treatment control arm)

ELIGIBILITY:
Inclusion Criteria:

* Cancer patient who has plan to receive first cycle of cisplatin >= 60 mg/m2
* Normal serum creatinine and creatinine clearance >= 50 ml/min
* Age < 75 years old
* Serum albumin >= 3 g/dl
* Plan to receive optimal antiemetic regimen consisting of olanzapine or neurokinase 1 receptor antagonist

Exclusion Criteria:

* The patient who receives other chemotherapy with adminstration volume higher than 500 ml
* Prior heart failure or known left ventricular ejection fraction > 50%
* Prior renal dysfunction within 3 months
* Uncontrolled renal disease
* current use of diuretic or non-steroidal anti-inflammatory drug (NSAIDs) or starting angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blockade (ARB) within 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-01-07 (Estimated); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
renal dysfunction at least grade 1 following cisplatin treatment in short hydration group | from starting cisplatin to 4-week after cisplatin discontinuation
  increased serum creatinine of 0.3 mg/dl or serum creatinine >= 1.5-2x upper normal limit

SECONDARY OUTCOMES:
renal dysfunction >= grade 2 following cisplatin treatment in short hydration group | from starting cisplatin to 4-week after cisplatin discontinuation
  serum creatinine > 2-3x upper normal limit
rate of cisplatin modification due to adverse effects in short hydration group | from starting cisplatin to 4-week after cisplatin discontinuation
  delay or dose reduction or discontinuation of cisplatin due to adverse effect

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jantarat A, Thamlikitkul L, Thephamongkhol K, Setakornnukul J, Phisalprapa P, Kositamongkol C, Srithongkul T, Ithimakin S. Efficacy and Safety of Short Intravenous Hydration for Preventing Nephrotoxicity From High-Dose Cisplatin: A Randomized, Open-Label, Phase II Trial. JCO Glob Oncol. 2025 Jan;11:e2400515. doi: 10.1200/GO-24-00515. Epub 2025 Jan 16. PMID 39819128